CLINICAL TRIAL: NCT01182285
Title: A Phase II Trial of Valproic Acid in Patients With Advanced Thyroid Cancers of Follicular Origin
Brief Title: A Phase II Trial of Valproic Acid in Patients With Advanced Thyroid Cancers of Follicular Cell Origin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100041; 10-C-0041
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Thyroid Neoplasm
Keywords: Depakote; Poorly Differentiated Thyroid Cancer; RAI Uptake; Thyrogen
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Valproic Acid; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A - Phase I Radioiodine-Resistant (Experimental): Drug: Valproic Acid Week 1 - 10 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening
  Interventions: Drug: Valproic Acid
- B1 - Phase 2 Schedule 1 (Active Comparator): Drug: Valproic Acid Week 11 - 17 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Drug: Cytomel (25 micrograms) Patients who exhibit an increased radioiodine uptake on Thyrogen scan post valproic acid therapy at week 10. Begin Liothyronine Sodium (Cytomel) for 4 weeks (25 micrograms twice a day)
  Interventions: Drug: Valproic Acid; Drug: Liothyronine Sodium
- B2 - Phase 2 Schedule 2 (Active Comparator): Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — Week 1:
  (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening
Drug: Liothyronine Sodium — Patients who exhibit an increased radioiodine uptake on Thyrogen scan post valproic acid therapy at week 10. Begin Cytomel for 4 weeks (25 micrograms twice a day)
  Other Names: Cytomel
  Arms: B1 - Phase 2 Schedule 1

SUMMARY:
Background:

* Patients who have advanced thyroid cancer have a low long-term survival rate. These types of thyroid cancer do not respond well to conventional surgery or radiation, or to specific thyroid cancer treatments such as radioactive iodine treatment and thyroid hormone for thyroid stimulating hormone (TSH) suppression.
* Valproic acid has long been approved as an anticonvulsant to treat seizures in patients with epilepsy. It has also been used to treat bipolar disorder. Recent studies have shown that valproic acid has promising effects in thyroid cancer treatment because it may help destroy cancer cells and help conventional treatments be more effective. However, valproic acid is not approved for thyroid cancer and is therefore an investigational drug.

Objectives:

* To determine whether valproic acid can inhibit tumor growth or induce tumor cell death.
* To determine whether valproic acid can make tumor cells increase their uptake of radioiodine.

Eligibility:

- Individuals at least 18 years of age who have advanced-stage thyroid cancer that is either unresponsive to conventional treatments or fails to absorb radioiodine.

Design:

* Eligible participants will continue on the standard thyroid hormone suppression therapy and begin receiving valproic acid for a total of 10 weeks. Participants will keep a study diary to record doses and side effects, and will have regular clinic visits to provide blood samples and receive additional valproic acid.
* After 10 weeks, participants will have a Thyrogen scan to measure radioiodine uptake after valproic acid therapy. Tumor biopsies and blood samples will be taken at this time.
* If there is increased radioiodine uptake on the scan, participants will have additional radioiodine therapy.
* If there is no increased uptake on the scan, participants will continue on valproic acid for 7 more weeks. After 16 total weeks of treatment, additional blood samples and scans will be taken. Participants may continue to take valproic acid if the thyroid cancer appears to be responding to the treatment.
* Follow-up visits will be scheduled at 3, 6, 9 (for patients continuing on valproic acid only), and 12 months.

DETAILED DESCRIPTION:
Background:

Patients who have advanced differentiated thyroid cancers (Stage IV) have a five-year survival of only 25%. Clinically this results in more aggressive growth, metastasis, decreased or loss of iodine uptake in the tumor, and tumors that may be refractory to conventional treatment: surgical resection, radioactive iodine treatment and thyroid hormone for Thyroid Stimulating Hormone (TSH) suppression.

In thyroid cancer, valproic acid, at clinically achievable concentrations, has an antiproliferative and differentiating effect.

We hypothesize that valproic acid may inhibit proliferation and induce differentiation in thyroid cancer cells so that 131-I may detect residual disease and be more effective for radioiodine ablation of thyroid cancer cells of follicular cell origin.

Objectives:

The primary goal of this study is to determine if valproic acid will have an antineoplastic and differentiation effect in patients with advanced and or metastatic thyroid cancer of follicular cell origin.

Eligibility:

Unresectable advanced and/or poorly differentiated thyroid cancers of follicular cell origin (excluding anaplastic and medullary thyroid cancer) that have no uptake (less than 1%) on radioiodine scan or are unresponsive to radioiodine therapy.

Elevated serum thyroglobulin (Tg) level (greater than 100ng/ml on thyroid hormone; greater than 10ng/ml off thyroid hormone).

Design:

This will be an open label phase II study to assess the efficacy of valproic acid therapy as an antiproliferative and differentiation agent in patients with incurable differentiated thyroid cancer (unresponsive and/or radioiodine negative and unresectable).

Oral valproic acid will be administered to reach a therapeutic serum level (50 to 100 microgram/ml).

The number of patients to be enrolled is 25 with an interim analysis of response once 13 patients are evaluable for response. It is anticipated that five patients may be enrolled per year.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Advanced/poorly differentiated thyroid cancers of follicular cell origin that have no uptake (less than 1%) on radioiodine scan or are unresponsive to radioiodine therapy. Unresponsiveness to radioiodine therapy is defined as a patient s thyroglobulin not falling to less than 2ng/ml within 6 months after previous radioiodine ablative treatment.
  2. Extensive (invasive) loco-regional tumor mass and/or metastatic spread, rendering patient inoperable.
  3. Thyroglobulin (Tg) levels greater than or equal to 100 ng/ml in the absence of Tg antibodies. Patients who are Tg-antibody (Tg-Ab) positive may be included despite a lower Tg level if they have detectable disease on cross sectional imaging. (The presence of Tg-Ab may lead to falsely low Tg levels and therefore render the Tg a less sensitive marker of disease. However, Tg-Ab has been shown to also act as a tumor marker, and will be used as an endpoint for the study in patients who are Tg-Ab positive.).
  4. Within 18 months of enrollment, patients must have had an radioactive iodine (RAI) scan, showing no or therapeutically insignificant RAI uptake (less than or equal to 1%).
  5. Initial therapy must have included total/near-total thyroidectomy and RAI ablation therapy.
  6. Patients must have had no chemotherapy, radiotherapy, or biologic therapy for their malignancy in the month prior to treatment and must have recovered from all side effects of therapeutic and diagnostic interventions.
  7. Greater than or equal to 18 years of age.
  8. Must be able to understand and sign the Informed Consent Document.
  9. Clinical performance status of Eastern Oncology Cooperative Group (ECOG) less than or equal to 1.
  10. Life expectancy of greater than three months.
  11. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (HCG) within 72 hours prior to study entry and must be willing to practice effective birth control to prevent pregnancy while receiving treatment and for three months after treatment is discontinued. All males of child fathering potential must also be willing to practice effective birth control.
  12. Laboratory results must be within the following parameters before entry:
* Absolute Neutrophil Count greater than 750 cells/mm(3)
* Hemoglobin greater than 8.0 gm/dl
* Platelet count greater than 75000/mm(3)
* Creatinine less tha 1.5 times upper limit of normal (ULN)
* Total protein greater than 6.4.
* Total bilirubin should be less than 1.5 times ULN.
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic (SGOT), alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) less than 1.5 times ULN.
* Amylase less than 1.5 times ULN
* Ammonia less than 1.5 times ULN

EXCLUSION CRITERIA:

1. Allergy to valproic acid.
2. Current coexisting malignancy other than basal cell carcinoma.
3. Women of child-bearing potential who are pregnant or breastfeeding.

   Valproic acid is a known teratogen, causing primary neural tube defects, facial abnormalities, and skeletal malformation; therefore pregnant women will be excluded. Additionally, patients that become pregnant while on study protocol will be discontinued immediately.
4. Active systemic infections, coagulation disorders or other major medical illnesses.
5. Patients taking tolbutamide, warfarin, zidovudine, benzodiazepines, clonazepam, diazepam.
6. Seizure disorder.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09-24 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies L, Welch HG. Increasing incidence of thyroid cancer in the United States, 1973-2002. JAMA. 2006 May 10;295(18):2164-7. doi: 10.1001/jama.295.18.2164. PMID 16684987
- [Background] Hundahl SA, Fleming ID, Fremgen AM, Menck HR. A National Cancer Data Base report on 53,856 cases of thyroid carcinoma treated in the U.S., 1985-1995 [see commetns]. Cancer. 1998 Dec 15;83(12):2638-48. doi: 10.1002/(sici)1097-0142(19981215)83:123.0.co;2-1. PMID 9874472
- [Background] Goretzki PE, Simon D, Frilling A, Witte J, Reiners C, Grussendorf M, Horster FA, Roher HD. Surgical reintervention for differentiated thyroid cancer. Br J Surg. 1993 Aug;80(8):1009-12. doi: 10.1002/bjs.1800800826. PMID 8402050
- [Result] Nilubol N, Merkel R, Yang L, Patel D, Reynolds JC, Sadowski SM, Neychev V, Kebebew E. A phase II trial of valproic acid in patients with advanced, radioiodine-resistant thyroid cancers of follicular cell origin. Clin Endocrinol (Oxf). 2017 Jan;86(1):128-133. doi: 10.1111/cen.13154. Epub 2016 Sep 8. PMID 27392538

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five and eight participants were enrolled from University of California San Francisco (UCSF) and the National Institutes of Health (NIH), respectively.
Groups:
- A - Phase 1 Radioiodine Resistant Thyroid Cancer: Drug: Valproic Acid Week 1 - 10 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening
- B1 - Phase 2 Schedule 1 (Increased Radioiodine Uptake): Drug: Valproic Acid Week 11 - 17 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Drug: Cytomel (25 micrograms) Patients who exhibit an increased radioiodine uptake on Thyrogen scan post valproic acid therapy at week 10. Begin Liothyronine Sodium (Cytomel) for 4 weeks (25 micrograms twice a day)
- B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake): Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by RECIST criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
Period: First Intervention Week 1-10
Arm/Group | A - Phase 1 Radioiodine Resistant Thyroid Cancer | B1 - Phase 2 Schedule 1 (Increased Radioiodine Uptake) | B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake)
Started | 13 | 0 | 0
Completed | 10 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0
Period: Second Intervention Week 11-17
Arm/Group | A - Phase 1 Radioiodine Resistant Thyroid Cancer | B1 - Phase 2 Schedule 1 (Increased Radioiodine Uptake) | B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake)
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Third Intervention Week 11-52
Arm/Group | A - Phase 1 Radioiodine Resistant Thyroid Cancer | B1 - Phase 2 Schedule 1 (Increased Radioiodine Uptake) | B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake)
Started | 0 | 0 | 8 (2 subj. taken off study after completing ph 1: 1 due to a negative uptake scan & one off due to PD.)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 8
Not completed — Disease Progression | 0 | 0 | 6
Not completed — Other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Five and eight participants were enrolled from University of California San Francisco (UCSF), and the National Institutes of Health, respectively.
Groups:
- All Participants (Phase 1 and Phase 2 Schedule 2): A- Phase 1 Radioiodine-Resistant Drug: Valproic Acid Week 1 - 10 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening
  B2 - Phase 2 Schedule 2 Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by RECIST criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
Arm/Group | All Participants (Phase 1 and Phase 2 Schedule 2)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.08 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: RAI (Radioactive Iodine) Uptake and Tg (Thyroglobulin) Level Compared Pre and Post- Valproic Treatment
Description: Complete response (CR) is increased Rai uptake on post- valproic acid therapy at week 10, AND a decrease in Tg level to less than 2 ng/ml (or a decrease in Tg-Ab level to less than 2.0 IU/ml) at 10 weeks AND disappearance of all lesions at 16 weeks. Partial response (PR) is increased Rai uptake on post-valproic scan at week 10, OR a decreased Tg level (or a decrease in Tg Ab (Tg antibody) level by more than 20%) at 10 weeks AND 30% decrease in target lesion at 16 weeks. Stable disease (SD) is no change in RAI uptake AND Tg levels (or TG-Ab level) AND no significant change of lesions at 16 weeks. Progressive disease (PD) is tumor mass increases OR Tg levels (or Tg-Ab levels) increases over 10 weeks OR at least 20% increase in target lesion at 16 weeks.
Time Frame: Entry to study and after 10 weeks of treatment for Phase 1, and 10 weeks of treatment to 16 weeks of treatment for phase 2.
Population: 13 participants were enrolled in phase 1 and 8/13 (5 from University of California San Francisco (UCSF) moved on from phase 1 to the phase 2 schedule 2 portion. However, Tg data from UCSF is unavailable for 5 of the participant, thus only 3 were analyzed in the phase 2 portion.
Measure: Count of Participants; unit: Participants
Arm/Group | A - Phase 1 Radioiodine Resistant Thyroid Cancer | B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake)
Number analyzed (Participants) | 13 | 3
Participants
  Tg start - >900 ng/ml | 6 | 1
  Tg start - 707 ng/ml | 1 | 0
  Tg start - 661 ng/ml | 1 | 0
  Tg start - 362 ng/ml | 0 | 1
  Tg start - 289 ng/ml | 1 | 0
  Tg start - 183 ng/ml | 0 | 1
  Tg start - 154 ng/ml | 1 | 0
  Tg start - 101 ng/ml | 1 | 0
  Tg start - 99 ng/ml | 1 | 0
  Tg start - 15.7 ng/ml | 1 | 0
  antiTg start - 142 IU/ml | 1 | 0
  antiTg start - 220 IU/ml | 0 | 1
  antiTg start - <20 IU/ml | 7 | 2
  Tg end - >900 ng/ml | 4 | 1
  Tg end - 749 ng/ml | 1 | 0
  Tg end - 702 ng/ml | 1 | 0
  Tg end - 630 ng/ml | 1 | 0
  Tg end - 480 ng/ml | 1 | 1
  Tg end - 362 ng/ml | 0 | 0
  Tg end - 204 ng/ml | 1 | 0
  Tg end - 184 ng/ml | 0 | 1
  Tg end - 183 ng/ml | 0 | 0
  Tg end - 128 ng/ml | 1 | 0
  Tg end - 61 ng/ml | 1 | 0
  Tg end - 10.8 ng/ml | 1 | 0
  Tg end - none | 1 | 0
  antiTg end - 338 IU/ml | 1 | 0
  anti Tg end - 220 IU/ml | 0 | 0
  antiTg end - 83 IU/ml | 1 | 0
  antiTg end - 80 IU/ml | 0 | 1
  anti Tg end - <20 IU/ml | 5 | 2
  antiTg end - none | 1 | 0
  RAI uptake pre-treatment - none | 13 | 0
  RAI uptake post treatment - none | 10 | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 41 months and 11 days
Population: Adverse events are not reported per Arm. All adverse events were reported to include phases 1 and 2 since it is analyzed throughout the whole study.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: A - Phase 1 Radioiodine Resistant Thyroid Cancer Drug: Valproic Acid Week 1 - 10 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake) Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by RECIST criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 13
Participants | 8

3. Secondary Outcome: Best Overall Response
Description: Best overall response was assessed by radioiodine uptake. Complete response (CR) is increased Rai (radioiodine) uptake on post- valproic acid therapy at week 10, AND a decrease in Tg (thyroglobulin ) level to less than 2 ng/ml (or a decrease in Tg-Ab (thyroglobulin antibodies) level to less than 2.0 IU/ml) at 10 weeks AND disappearance of all lesions at 16 weeks. Partial response (PR) is increased Rai uptake on post-valproic scan at week 10, OR a decreased Tg level (or a decrease in Tg Ab (Tg antibody) level by more than 20%) at 10 weeks AND 30% decrease in target lesion at 16 weeks. Stable disease (SD) is no change in RAI uptake AND Tg levels (or TG-Ab level) AND no significant change of lesions at 16 weeks. Progressive disease (PD) is tumor mass increases OR Tg levels (or Tg-Ab levels) increases over 10 weeks OR at least 20% increase in target lesion at 16 weeks.
Time Frame: Week 16
Population: Best overall response was not assessed for the phase 1 portion.
Measure: Count of Participants; unit: Participants
Groups:
- B2 - Phase 2 Schedule 2 (No Increased Radiiodine Uptake): Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by RECIST criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
Arm/Group | B2 - Phase 2 Schedule 2 (No Increased Radiiodine Uptake)
Number analyzed (Participants) | 8
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 6
  Unknown | 1

4. Secondary Outcome: NIS (Na/I-symporter) Expression
Description: NIS (Na/I-symporter) Expression is assessed by quantitative reverse transcription (RT) polymerase chain reaction (PCR) and immunohistochemistry (IHC). NIS mRNA expression was measured by quantitative RT PCR from biopsy samples.
Time Frame: Entry to study and after 10 weeks of treatment
Population: There is no standard of error to report. The acronym GAPDH expanded is glyceraldehyde 3-phosphate dehydrogenase. Only 1 participant was analyzed because biopsies were not performed in 12 subjects.
Measure: Median (Standard Error); unit: percent expression
Arm/Group | A - Phase 1 Radioiodine Resistant Thyroid Cancer
Number analyzed (Participants) | 1
percent expression
  Pre-treatment NIS expression (relative to GAPDH) | 21 (0)
  Post-treatment NIS expression (relative to GAPDH) | 25 (0)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 41 months and 11 days
Description: Adverse events are not reported per Arm. All adverse events were reported to include phases 1 and 2 since it is analyzed throughout the whole study. No adverse events were recorded for participants at University of California San Francisco (UCSF).
Groups:
- All Participants (Phase 1 and Phase 2 Schedule 2): A - Phase 1 Radioiodine Resistant Thyroid Cancer Drug: Valproic Acid Week 1 - 10 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening B2 - Phase 2 Schedule 2 (No Increased Radioiodine Uptake) Drug: Valproic Acid Week 11 - 52 (Days 1-3): Valproic acid - 500 mg every evening (Day 4-7): Valproic acid - 500 mg twice daily (morning and evening) Weeks 2 through 10: Valproic acid 500 mg every morning and 1000 mg every evening Weeks 17-52: Patients who show a response by RECIST criteria or have a decreased thyroglobulin level from Day 1 of the treatment (registered as a partial response to the treatment) will continue on valproic acid at their current dose for a total of 52 weeks.
Arm/Group | All Participants (Phase 1 and Phase 2 Schedule 2)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (Phase 1 and Phase 2 Schedule 2) (N=13)
Confusion (Psychiatric disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (Phase 1 and Phase 2 Schedule 2) (N=13)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (8)
Platelet count decreased (Investigations) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT01182285/Prot_ICF_000.pdf